CLINICAL TRIAL: NCT02040064
Title: Phase I, Open-label, Safety, Tolerability and Preliminary Efficacy Study of Tremelimumab in Combination With Gefitinib in EGFR Mutant NSCLC Patients
Brief Title: Tolerability and Efficacy of Tremelimumab in Combination With Gefitinib in NSCLC Patients
Acronym: GEFTREM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-003015-21; 2013/2028 (Other: CSET number)
Record Dates: First submitted 2014-01-10; First posted 2014-01-20 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): * Cohort 1: Tremelimumab 3 mg/kg every 4 Weeks plus Gefitinib 250 mg/daily, 6 patients (+ 6 patients if 3 mg/kg is the MTD)
  * Cohort 2: Tremelimumab 6 mg/kg every 4 Weeks plus Gefitinib 250 mg/daily, 6 patients (+ 6 patients if 6 mg/kg is the MTD)
  * Cohort 3: Tremelimumab 10 mg/kg every 4 Weeks plus Gefitinib 250 mg/daily, 6 patients (+ 6 patients if 10 mg/kg is the MTD)
  Interventions: Drug: Gefitinib; Drug: Tremelimumab

INTERVENTIONS:
Drug: Gefitinib — Oral tablet
Drug: Tremelimumab — IV

SUMMARY:
This is an open-label phase 1, safety, PK, and preliminary efficacy study of oral Gefitinib and IV Tremelimumab in previously treated NSCLC patients who have documented evidence of an activating mutation in the EGFR gene and have failed treatment with an EGFR inhibitor such as Erlotinib or Gefitinib. The primary objective of this phase I, is to determine the safety and tolerability of oral Gefitinib in combination with escalating doses of Tremelimumab and to establish a recommended phase 2 dose. Secondary objectives include evaluation of, pharmacokinetics, immunogenicity, antitumor activity of Gefitinib and Tremelimumab combination. The exploratory objectives are to evaluate biomarkers that may correlate with activity or prospectively identify patients likely to respond to Tremelimumab and Gefitinib.

The biological rationale for such a study is that even though the disease is progressing it is likely that EGFR sensitive clones, although diminished under the pressure from the EGFR TKI, are still present. Therefore, withdrawing the inhibitory pressure of the EGFR TKI can potentially allow regrowth of the EGFR sensitive cells. On the other hand, the proliferation of EGFR resistant clones needs to be suppressed by another therapeutic approach. Until today no association of chemotherapy and TKI EGFR has demonstrated clinical benefit. Moreover, patients may have received chemotherapy and the likelihood of chemosensitivity is very low. So, the association of Gefitinib with immune checkpoint blockade is very attractive and may result in clinical benefit in NSCLC with EGFRmut.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent ;
2. Female or male patients aged 18 years or over at the time of consent ;
3. World Health Organisation (WHO) Performance Status 0 to 1 (Appendix C) ;
4. Cytologically or histologically confirmed NSCLC with an activating EGFR TK mutations known to be associated with EGFR TKI sensitivity (i.e., G719X, exon 19 deletion, L858R, L861Q) as determined locally using a well-validated and robust methodology ;
5. Prior objective clinical benefit defined by either partial, complete or SD (>/= 4months) after initiation of EGFR TKI treatment ;
6. Patients could have received first line chemotherapy or chemotherapy between the EGFR TKI and inclusion in the study but must present a systemic objective progression ;
7. A washout period is not required for patients who are being treated with Gefitinib at the time of study entry. A washout period of at least 14 days is required for patients being treated with an irreversible EGFR TKI, chemotherapy, of at least 5 days for patients being treated with Erlotinib and at least five half-life for other treatments ;
8. Locally advanced Stage IIIB not suitable for local therapy of curative intent or Stage IV (metastatic) disease ;
9. At least one lesion, not previously irradiated and not chosen for fresh biopsy during the study screening period, that can be accurately measured at baseline as >/= 10mm in the longest diameter (except lymph nodes which must have short access >/= 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements ;
10. No standard therapy is considered appropriate. Prior treatment with chemotherapy is not mandated if either the patient refuses treatment with chemotherapy, or if, in the opinion of the investigator it is acceptable to delay treatment with chemotherapy ;
11. Recovered from all toxicities associated with prior treatment, to acceptable baseline status, or a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade of 0 or 1, except for toxicities not considered a safety risk, such as alopecia or vitiligo ;
12. Adequate bone marrow, hepatic, and renal function determined within 14 days prior to enrollment defined as:

    1. Platelet count >/= 100,000/mm3
    2. Absolute neutrophil count >/= 1,500/mm3
    3. Haemoglobin >/= 9 g/dL
    4. Total bilirubin </= 1.5 × ULN (upper limit of normal)
    5. Aspartate transaminase (AST) and alanine transaminase (ALT) </= 2.5 × ULN
    6. Creatinine </=1.5 times ULN concurrent with creatinine clearance >/= 50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
13. Negative screening test results for human immunodeficiency virus (HIV), hepatitis A, B and C. If positive results are not indicative of true active or chronic infection, the subjects can enter the study ;
14. Negative pregnancy test in women of childbearing potential within 14 days prior to treatment initiation. Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 6 months after the final dose of investigational product. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Day 1 through 90 post last dose ; For inclusion in the optional genetic component of the study, subjects must fulfill the following additional criterion:
15. Provide signed, written, and dated informed consent for genetic research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent.

Exclusion Criteria:

1. Known severe hypersensitivity to Gefitinib or any of the excipients of the product ;
2. Previous EGFR TKI toxicity requiring discontinuation of treatment with the EGFR TKI (> 4 weeks), or considered, by the investigator, to be difficult to manage ;
3. Prior treatment with monoclonal antibody against CTLA-4, programmed cell death 1 (PD1) or programmed cell death 1 ligand 1 (PD-L1) ;
4. Prior surgery or radiotherapy is allowed if completed more than 6 months before start of study treatment. Palliative radiotherapy must be completed at least 2 weeks before start of study treatment with no persistent radiation toxicity ;
5. Considered to require radiotherapy to the lung at the time of study entry or in the near future ;
6. Spinal cord compression or brain metastases unless asymptomatic, treated and stable, and not requiring steroids for at least 2 weeks prior to the start of study treatment ;
7. Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease ;
8. Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline ;
9. Insufficient lung function as determined by either clinical examination or an arterial oxygen tension (PaO2) of < 70 Torr ;
10. Females who are pregnant or breastfeeding ;
11. History of chronic inflammatory or autoimmune disease (eg Addison's disease, multiple sclerosis, Graves' disease, Hashimoto's thyroiditis, rheumatoid arthritis, hypophysitis, etc) with symptomatic disease within the last 3 years prior to study entry. Note: Active vitiligo or a history of vitiligo is not a basis for exclusion ;
12. Any serious uncontrolled medical disorder or active infection that would impair the subject's ability to receive investigational product, such as conditions associated with frequent diarrhoea ;
13. Clinically relevant cardiovascular disease, i.e., myocardial infarction or other severe coronary artery diseases within the prior 6 months, cardiac arrythmia requiring medication, uncontrolled hypertension, overt cardiac failure or not compensated chronic heart disease in NYHA class II or more ;
14. Active or history of, diverticulitis. Note that diverticulosis is permitted ;
15. Active or history of, inflammatory bowel disease (eg, colitis, Crohn's), irritable bowel disease, coeliac disease or other serious gastrointestinal chronic conditions associated with diarrhea ;
16. Active, or history of, systemic lupus erythematosis or Wegener's granulomatosis ;
17. History of sarcoidosis syndrome ;
18. Currently receiving systemic corticosteroids or other immunosuppressive medications, or has a medical condition that requires the chronic use of corticosteroids. Inhaled and topical steroids are permitted ;
19. Vaccination with a live attenuated vaccine within one month prior to starting study treatment ;
20. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study ;
21. History of other malignancy unless the subject has been disease-free for at least 2 years. Noninvasive cancer history (such as carcinoma in situ [CIS] that has been resected) is allowed ;
22. Any condition that would prohibit the understanding or rendering of information and consent and compliance with the requirements of this protocol ;
23. Enrolment in another clinical study (except observational studies) ;
24. Previous enrolment or treatment in the present study ;
25. In addition, the following are considered criteria for exclusion from the genetic research:

    * Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.
    * Previous allogenic bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of the association between Gefitinib (fixed dose) and Tremelimumab (dose escalation) | Up to 42 days
  The primary objective of this phase 1 study is to determine the safety and tolerability of oral Gefitinib in combination with three escalating doses of Tremelimumab and to establish a recommended phase 2 dose. Overall safety profile will be characterized by type, frequency, severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCICTCAE] Version 4.03), timing of adverse events and laboratory abnormalities in the first and in the following cycles

SECONDARY OUTCOMES:
Anti-tumour activity of Gefitinib + Tremelimumab | From day 1 cycle 1 every 8 weeks for 24 weeks and then every 6 weeks until progression or death whichever comes first assessed up to 30 months
  To obtain a preliminary assessment of the anti-tumour activity of Gefitinib + Tremelimumab by evaluation of tumour response using modified Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 and evaluation of Disease control rate and PFS
Immunogenicity of Tremelimumab in combination with Gefitinib | At day 1 cycle 1 and then every 8 weeks from day 1 cycle 2 until progression or death whichever comes first assessed up to 30 months
  Immunogenicity results will be analyzed descriptively by summarizing the number and percentage of subjects who develop detectable anti-Tremelimumab antibodies. The immunogenicity titer will be reported for samples confirmed positive for the presence of anti-Tremelimumab antibodies.
Pharmacokinetics of Gefitinib | At first Tremelimumab administration and then every 4 weeks until progression or death whichever comes first assessed up to 30 months
  Gefitinib pharmacokinetic parameters comprise the area under the curve from time t0 to t (AUC0-t), AUC from time t0 to the infini (AUC0-∞) and maximal concentration (Cmax)
Pharmacokinetics of Tremelimumab | Before and after injection of Tremelimumab at day 1 cycle 1 and at day 8 and day 15 of cycle 1 and then before and after injection at day 1 for every cycle (4 weeks) until progression or death whichever comes first assessed up to 30 months
  Tremelimumab pharmacokinetic parameters comprise the area under the curve from time t0 to t (AUC0-t), AUC from time t0 to the infini (AUC0-∞) and maximal concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: David Planchard, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Riudavets M, Naigeon M, Texier M, Dorta M, Barlesi F, Mazieres J, Varga A, Cassard L, Boselli L, Grivel J, NgoCamus M, Lacroix L, Mezquita L, Besse B, Chaput N, Planchard D. Gefitinib plus tremelimumab combination in refractory non-small cell lung cancer patients harbouring EGFR mutations: The GEFTREM phase I trial. Lung Cancer. 2022 Apr;166:255-264. doi: 10.1016/j.lungcan.2021.11.018. Epub 2021 Dec 3. PMID 34953624